CLINICAL TRIAL: NCT02396056
Title: Enhanced Guided Bone Regeneration in Localized Osseous Alveolar Defects by Using a Novel Perforated Resorbable Barrier Membrane
Brief Title: Enhancing Guided Bone Regeneration by Modifying a Resorbable Membrane
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StonyBrookU
Record Dates: First submitted 2015-03-18; First posted 2015-03-24 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Alveolar Ridge Augmentation
Keywords: Guided Bone Regeneration; Gingival Mesenchymal Stem Cells

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Occlusive Membrane (OM) (Sham Comparator): Five patients will be randomly assigned to the OM group.
  Interventions: Other: BioMend Extend
- Modified Perforated Membrane (MPM) (Experimental): Five patients will be randomly assigned to the MPM group.
  Interventions: Other: Modified BioMend Extend

INTERVENTIONS:
Other: BioMend Extend — Biomend Extend is a resorbable collagen membrane used for guided tissue and bone regeneration.
  Arms: Occlusive Membrane (OM)
Other: Modified BioMend Extend — Biomend Extend is a resorbable collagen membrane used for guided tissue and bone regeneration. This membrane will be perforated to allow the passage of cells and growth factors that can potentially enhanced bone augmentation.
  Arms: Modified Perforated Membrane (MPM)

SUMMARY:
Guided bone regeneration (GBR) procedures have significantly evolved over the last 20 years. Significant advances have been made with various barrier membranes with or without the use of bone grafts and other materials. Some of the main limitations of non-resorbable barriers included cytotoxicity and need for removal, which can adversely affect the regenerated bone volume. Similar GBR success has been documented extensively with cell occlusive resorbable barriers membranes. Recently, the investigators demonstrated supracrestal bone regeneration in guided tissue regeneration procedures in humans with the use of novel perforated barrier membrane (MPM). The perforation allows mesenchymal stem cells and other progenitor cells present in the gingival tissues to migrate into the osseous defect and contribute to the osseous regeneration potential.

The objective of this study is to investigate the GBR potential of MPM in alveolar ridge defects, relative to a similar occlusive barrier. Ten non-smoking patients that need localized alveolar ridge augmentation prior to implant placement will be included into the study. Patients will be divided into two groups, as follows: occlusive bovine collagen membrane (OM control group, 5 patients) and modified bovine perforated collagen membrane (MPM test group, 5 patients). All sites will be grafted with mineralized cortical bone allograft and when needed cortical bone pins will be use for site stability. A Cone Bean (CT) will be obtained prior to surgery and 6-8 months post treatment from which volumetric width changes will be quantify. A bone biopsy will be obtained at the time of implant placement (~6-8 months) to determine residual graft particles and new bone formation. Dimensional width changes will be assess at 6-8 months during re-entry for implant placement. Soft tissue healing will be assessed at 2, 4, 8, 16 weeks and 6 months.

This study can potentially impact current bone augmentation techniques and may lead to the modification of existing commercial membranes that will enhance site development prior to implant placement. The contribution of progenitor cells to the osseous defect might lead to greater bone formation and possible faster wound healing.

ELIGIBILITY:
Inclusion Criteria:

* at the augmentation site, the alveolar ridge must be deficient in a buccolingual dimension (< 5.5 mm): Class 1 Seibert defects.
* alveolar ridges to be augmented must have a minimum of 4 mm of keratinized gingiva extending the length of the planned augmentation.

Exclusion Criteria:

* general contraindications to implant surgery
* subjected to irradiation, chemotherapy or immunosuppressive therapy over the past 5 years
* poor oral hygiene and motivation
* uncontrolled diabetes
* pregnant or lactating
* substance abusers
* current smokers
* psychiatric problems or unrealistic expectations
* acute infection in the area intended for implant placement
* positive to HIV and hepatitis B and C
* affected by autoimmune diseases such as arthritis rheumatoid, systemic lupus erythematosus, sclerodermia, Sjo ̈gren syndrome and dermatomyositis polymyositis
* treated or under treatment with intravenous amino-bisphosphonates
* subjected previously to reconstructive procedures of the posterior mandible and
* under chronic treatment with steroids or non-steroidal anti-inflammatory drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Clinical horizontal bone augmentation results through direct measurement. | at 6 months post treatment

SECONDARY OUTCOMES:
Volumetric measurements with CBCT | pre- and 6 months post treatment

OTHER OUTCOMES:
De novo bone formation, and residual graft particles quantification with histomorphometric analysis | at 6 months post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine of Stony Brook University, Stony Brook, New York, United States